CLINICAL TRIAL: NCT00897728
Title: Colon and Breast Cancer Diagnostics. Clinical Protocol Associated With Cancer of the Breast.
Brief Title: Study of Tumor and Blood Samples From Women With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Curie (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000599189; CLCC-IC-COBRED-SEIN; CLCC-IC-2007-11; CLCC-RECF0632
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; HER2-positive breast cancer; triple-negative breast cancer; estrogen receptor-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at tumor and blood samples from women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess relapse locally or remotely using biomarkers collected from primary tumor and blood samples from women with breast cancer during the first 2 years after diagnosis.

Secondary

* Evaluate all relapses.
* Assess survival without relapse.
* Determine correlation between biomarkers and relapse.

OUTLINE: Primary tumor and blood samples collected during usual care of patients during the first 2 years after diagnosis are analyzed for biomarkers useful in monitoring and diagnosing breast cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of infiltrating unilateral breast cancer

  * No in situ disease (ductal or lobular)
  * No invasive bilateral synchronous disease
* Breast cancer at high risk, defined by at least 2 of the following factors:

  * Hormone receptor negative (HR-)
  * Axillary node positive
  * Histopathologic grade III
  * High mitotic index (as defined by the Curie Institute as > 20 mitoses per 10 high-power fields [HPF])
  * Tumor size ≥ 2 cm
  * HER2-positive (3 + IHC or FISH/ICHS positive)
  * Triple-negative tumors (HR- and HER2-negative)
* Initial thoracic-abdomino-pelvic and bone scans must be negative
* Underwent initial surgery

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Serum calcium normal (15.3 mg/dL) or normalized within 8 weeks after surgery
* No other invasive cancer within the past 5 years
* Not pregnant or nursing
* No psychological, familial, social, or geographical reasons that make monitoring impossible

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Local or remote relapse as assessed by biomarkers in tissue and blood samples collected during the first 2 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Henri Cottu, Study Chair — Institut Curie
Locations (1):
- Institut Curie Hopital, Paris, France